CLINICAL TRIAL: NCT00047164
Title: A Pilot Study of Ipilimumab (MDX-CTLA4, MDX-010) in Lymphoma
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Lymphoma or Colon Cancer That Has Not Responded to Vaccine Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Edward Janik, NCI - Metabolism Branch;MET
Masking: None | Purpose: Treatment
Other Study IDs: 020284; 02-C-0284; NCI-5744; CDR0000257563
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; recurrent adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage II adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II adult T-cell leukemia/lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Hodgkin Disease; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — Ipilimumab

INTERVENTIONS:
Biological: ipilimumab

SUMMARY:
RATIONALE: Monoclonal antibodies such as anti-cytotoxic T-lymphocyte-associated antigen-4 can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: This phase II trial is studying anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody to see how well it works in treating patients with lymphoma or colon cancer that has not responded to vaccine therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody in patients with follicular or mantle cell lymphoma, colon cancer, or prostate cancer refractory to vaccine therapy. (part I) (prostate cancer and mantle cell lymphoma closed to accrual as of 3/10/2005; colon cancer closed to accrual as of 9/28/05)
* Determine the toxicity of this drug at escalating doses in patients with follicular lymphoma. (part II)
* Determine the toxicity of this drug at escalating doses in patients with non-Hodgkin's lymphoma or Hodgkin's lymphoma. (part III)

Secondary

* Determine the ability of this drug to increase tumor-specific T-cell responses in these patients.
* Determine the ability of this drug to produce clinical tumor response in these patients.
* Determine the effect of this drug on suppressor T-cell populations (CD4+ and CD25+ cells) in these patients.

OUTLINE: This is a pilot, partial dose-escalation study.

* Part I (patients with prostate or colon cancer or follicular or mantle cell lymphomas) (prostate cancer and mantle cell lymphoma closed to accrual as of 3/10/2005; colon cancer closed to accrual as of 9/28/05): Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-CTLA4) IV over 90 minutes on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Part II (dose-escalation) (patients with follicular lymphomas only): Patients receive MDX-CTLA4 as in part I. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of MDX-CTLA4 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

* Part III (dose-escalation*) (patients with non-Hodgkin's or Hodgkin's lymphoma): Patients receive MDX-CTLA4 as in part II.

NOTE: No dose-escalation for lymphoma patients who have previously been treated with an allogeneic stem cell transplantation.

Patients are followed every other month.

PROJECTED ACCRUAL: A total of 89 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer (closed to accrual as of 3/9/2005)

  * Prior therapy on protocol NCI-00-C-0137 or NCI-00-C-0154
  * Progressive disease (2 consecutively rising PSA levels, new bone scan lesion, or progression of soft tissue)
  * PSA at least 5 ng/mL
  * Progressive androgen-independent disease

    * Disease progression at least 4 weeks after flutamide withdrawal OR
    * Disease progression at least 6 weeks after bicalutamide or nilutamide withdrawal OR
* Histologically confirmed follicular or mantle cell non-Hodgkin's lymphoma (mantle cell lymphoma closed to accrual as of 3/9/2005)

  * Prior therapy on protocol NCI-00-C-0133, NCI-01-C-0169, or NCI-00-C-0050
  * Progressive disease after standard treatment
  * Relapsed disease OR
* Histologically confirmed colon cancer (colon cancer closed to accrual as of 9/28/05)

  * Prior therapy on protocol NCI-99-C-0023
  * Progressive disease OR
* Histologically confirmed non-Hodgkin's lymphoma or Hodgkin's lymphoma

  * Progressive disease after standard treatment
  * No curative therapy exists
  * Prior allogeneic stem cell transplantation from a matched sibling or matched unrelated donor for an aggressive lymphoma allowed

    * Last infusion of allogeneic cells (either hematopoietic stem cells or donor lymphocytes) must have occurred > 90 days prior to study enrollment
* No other standard therapy available or refused such therapy
* No symptomatic or rapidly progressive malignancy requiring therapy
* No symptomatic CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* More than 2 months

Hematopoietic

* WBC at least 2,500/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 50,000/mm^3
* Hemoglobin at least 10 g/dL
* Hematocrit at least 30%

Hepatic

* Bilirubin no greater than 3.0 mg/dL (unless due to Gilbert's disease)
* SGOT and SGPT no greater than 3 times upper limit of normal
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine no greater than 2.0 mg/dL

Immunologic

* HIV negative
* Rheumatoid factor negative if history or evidence of arthritis
* Anti-nuclear antibody (ANA) titer no greater than 1:80 if history or clinical signs or symptoms of connective tissue disease
* No prior or active autoimmune disease (e.g., uveitis, rheumatoid arthritis, lupus erythematosus, autoimmune hemolytic anemia, ulcerative and hemorrhagic colitis, endocrine disorders [e.g., thyroiditis, hyperthyroidism, hypothyroidism, autoimmune hypophysitis/hypopituitarism, or adrenal insufficiency], sarcoid granuloma, myasthenia gravis, polymyositis,or Guillain-Barre syndrome)
* No positive antibody titers to autoimmune diseases

  * Rheumatoid factor positive allowed unless ANA titer is greater than 1:80 and there is a history of or clinical signs or symptoms of connective tissue disease
* No active infection

Other

* No other active malignancy within the past 5 years except adequately treated squamous cell or basal cell skin cancer, carcinoma in situ of the cervix, or superficial bladder cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* Recovered from prior vaccine therapy
* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-CTLA4) for patients in part I of study

  * Patients in part II of study may have had up to 4 prior treatments with MDX-CTLA4
* No concurrent vaccine therapy
* No concurrent infliximab

Chemotherapy

* At least 4 weeks since prior cytotoxic chemotherapy
* No concurrent mercaptopurine, methotrexate, or cyclophosphamide

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior steroids
* No concurrent systemic, inhaled, or topical steroids

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* At least 4 weeks since prior major surgery

Other

* Prior intervening therapy for prostate cancer, non-Hodgkin's lymphoma or colon cancer allowed
* No other concurrent investigational therapy
* No other concurrent immunosuppressants (e.g., cyclosporine or its analog)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2002-09; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Toxicity after every 3 courses of treatment and every month for up to a year after completion of study treatment

SECONDARY OUTCOMES:
T-cell response after every 3 courses of treatment and every month for up to a year after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: John E. Janik, MD, Study Chair — NCI - Metabolism Branch;MET
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States